CLINICAL TRIAL: NCT01339403
Title: Hiv Infection, Antiretroviral Therapy Use And Other Predictors Of Selected Clinical Events In Kaiser Permanente
Brief Title: Kaiser Permanente HIV Cohort Study
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: Kaiser Permanente (Other); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4001105
Record Dates: First submitted 2011-03-16; First posted 2011-04-20 (Estimated); Results first posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV infected: No study specific intervention, non-interventional trial
  Interventions: Other: non-interventional trial
- HIV-uninfected: No study specific intervention, non-interventional trial
  Interventions: Other: non-interventional trial

INTERVENTIONS:
Other: non-interventional trial — No study specific intervention, non-interventional trial
  Groups: HIV infected
Other: non-interventional trial — No study specific intervention, non-interventional trial
  Groups: HIV-uninfected

SUMMARY:
Human Immunodeficiency Virus (HIV) infected patients in the Kaiser Permanente HIV registry wil be followed in the usual clinical care to estimate the rates of specified clinical events. The rates will be stratified by relevant characteristics like age, CD4 counts, HIV Viral Load (VL), HIV medication history. The rates in the HIV infected cohort wil be compared with the rates of these events in patients in the Kaiser Permanente database who are not infected with HIV.

DETAILED DESCRIPTION:
All HIV infected patients in the database will be included without any sampling. A random sample of non-HIV infected patients will be included as comparator.

ELIGIBILITY:
Inclusion Criteria:

HIV infection.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected patients in the HIV Registry of Kasier Permanente Northern and Southern California and a matched cohort of non-HIV infected patients in Kaiser Permanente
Sampling Method: Non-Probability Sample
Enrollment: 282368 (Actual)
Dates: Start 2009-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001105&StudyName=Kaiser%20Permanente%20HIV%20Cohort%20Study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants infected and uninfected with Human Immunodeficiency Virus (HIV) were recruited and analyzed retrospectively in the Kaiser Permanente HIV registry.
Groups:
- Cohort 1: HIV Infected: Participants who were diagnosed with HIV infection and received HIV care during January 1, 1996 through December 31, 2006 (574 weeks) with follow-up extended up to 31st December 2011 (up to 835 weeks).
- Cohort 2: HIV Uninfected: Participants who were not diagnosed with HIV infection during January 1, 1996 through December 31, 2006 (574 weeks) with follow-up extended up to 31st December 2011 (up to 835 weeks).
Period: Overall Study
Arm/Group | Cohort 1: HIV Infected | Cohort 2: HIV Uninfected
Started | 24768 | 257600
Completed | 24768 | 257600
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: HIV Infected | Cohort 2: HIV Uninfected | Total
Number analyzed (Participants) | 24768 | 257600 | 282368
Age, Customized [Number; unit: participants]
  Less than (<) 35 years | 6883 | 76826 | 83709
  Between 35 and 39 years | 4919 | 50657 | 55576
  Between 40 and 44 years | 4700 | 47564 | 52264
  Between 45 and 49 years | 3701 | 37184 | 40885
  Between 50 and 54 years | 2302 | 22942 | 25244
  Between 55 and 59 years | 1246 | 12199 | 13445
  Between 60 and 64 years | 613 | 6154 | 6767
  Greater than (>) 65 years | 404 | 4074 | 4478
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2306 | 24134 | 26440
  Male | 22462 | 233466 | 255928

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Malignancies
Description: Incidence rate of malignancies was calculated as the number of events divided by person-time. Only the first diagnosis of each event per participant was included.Person-time was calculated as the sum of all time contributed by each individual who were Kaiser Permanente (KP) member from the date of HIV care initiation at that institution or January 1, 1996 for KP Northern California(KPNC) and January 1, 2000 for KP Southern California(KPSC) if in care prior to this date. Malignancies included acquired immunodeficiency syndrome (AIDS)-defining malignancies and non-AIDS defining malignancies.AIDS-defining malignancies included invasive cervical cancer,invasive non-Hodgkin's lymphoma and kaposi's sarcoma;non-AIDS defining malignancies cancers ascertained from the KP cancer registries.Overall data for non-AIDS and AIDS defining malignancies, along with individual data for AIDS-defining malignancies was reported. Incidence rate was computed as the number of events per 100,000 person-years.
Time Frame: Up to Week 835
Population: Analysis population included all participants enrolled in the study.
Measure: Number; unit: malignancies per 100,000 person-years
Arm/Group | Cohort 1: HIV Infected | Cohort 2: HIV Uninfected
Number analyzed (Participants) | 24768 | 257600
malignancies per 100,000 person-years
  Kaposi's sarcoma | 513 | 3
  Invasive non-Hodgkin's lymphoma | 238 | 20
  Invasive cervical cancer | 25 | 7
  Non-AIDS-defining cancer | 633 | 384
  AIDS-defining cancer | 740 | 23
Statistical Analysis 1: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Kaposi's sarcoma: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 166.1, 95% CI 2-sided [123.4 to 223.5]
Statistical Analysis 2: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Invasive non-Hodgkin's lymphoma: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 12.1, 95% CI 2-sided [10.3 to 14.2]
Statistical Analysis 3: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Invasive cervical cancer: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p = 0.059, Poisson Regression; Rate ratio = 3.4, 95% CI 2-sided [1.0 to 12.3]
Statistical Analysis 4: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Non-AIDS-defining cancers: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 1.7, 95% CI 2-sided [1.5 to 1.8]
Statistical Analysis 5: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; AIDS-defining cancer: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate Ratio = 166.1, 95% CI 2-sided [123.4 to 223.5]

2. Primary Outcome: Incidence Rate of Myocardial Infarction and Ischemia
Description: Incidence rate of cardiovascular (CVS)events including myocardial infarction (MI) and ischemia was calculated as the number of events divided by person-time. Only the first diagnosis of each event per participant was included. Person-time was calculated as the sum of all time contributed by each individual who were KP member from the date of HIV care initiation at that institution or January 1, 1996 for KPNC and January 1, 2000 for KPSC if in care prior to this date. Incidence rate was computed as the number of events per 100,000 person-years.
Time Frame: Up to Week 835
Population: Analysis population included all participants enrolled in the study.
Measure: Number; unit: CVS events per 100,000 person-years
Arm/Group | Cohort 1: HIV Infected | Cohort 2: HIV Uninfected
Number analyzed (Participants) | 24768 | 257600
CVS events per 100,000 person-years | 435 | 313
Statistical Analysis 1: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 1.4, 95% CI 2-sided [1.3 to 1.5]

3. Primary Outcome: Incidence Rate of Acquired Immunodeficiency Syndrome (AIDS)-Defining Opportunistic Infections
Description: Incidence rate of AIDS-defining opportunistic infections (OI) was calculated as the number of events divided by person-time.Only the first diagnosis of each event per participant was included.Person-time was calculated as the sum of all time contributed by each individual who were KP member from the date of HIV care initiation at that institution or January 1,1996 for KPNC and January 1,2000 for KPSC if in care prior to this date.OI were those that occurred on immune-compromised participants.AIDS-defining infections included:wasting syndrome;pneumocystis jirovecii pneumonia;recurrent pneumonia;cytomegalovirus;HIV-related encephalopathy;esophageal candidiasis;mycobacterium avium complex;cryptococcosis;mycobacterium tuberculosis;progressive multifocal leukoencephalopathy;lung candidiasis;toxoplasmosis of brain;coccidiomycosis;histoplasmosis;recurrent salmonella septicemia;chronic isosporiasis;cryptosporidiosis.Incidence rate was computed as the number of events per 100,000 person-years.
Time Frame: Up to Week 835
Population: Analysis population included all participants enrolled in the study.
Measure: Number; unit: infections per 100,000 person-years
Arm/Group | Cohort 1: HIV Infected | Cohort 2: HIV Uninfected
Number analyzed (Participants) | 24768 | 257600
infections per 100,000 person-years
  Wasting syndrome | 1002 | 15
  Pneumocystis jirovecii pneumonia | 760 | 2
  Recurrent pneumonia | 640 | 74
  Cytomegalovirus | 440 | 5
  HIV-related Encephalopathy | 405 | NA — No participant in this arm was evaluated for HIV-related encephalopathy, since only HIV infected participants were assessed for this infection.
  Esophageal Candidiasis | 383 | 6
  Mycobacterium avium complex | 259 | 3
  Cryptococcosis | 187 | 1
  Mycobacterium tuberculosis | 157 | 25
  Progressive multifocal leukoencephalopathy | 78 | 0
  Lung Candidiasis | 63 | 6
  Toxoplasmosis of brain | 58 | 1
  Coccidiomycosis | 9 | 1
  Histoplasmosis | 20 | 2
  Recurrent Salmonella septicemia | 2 | 0
  Chronic Isosporiasis | 0 | 0
  Cryptosporidiosis | 72 | 0
Statistical Analysis 1: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Wasting syndrome: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 65.7, 95% CI 2-sided [57.1 to 75.7]
Statistical Analysis 2: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Pneumocystis jirovecii pneumonia: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 428.5, 95% CI 2-sided [292.2 to 628.5]
Statistical Analysis 3: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Pneumonia, recurrent: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 8.7, 95% CI 2-sided [7.9 to 9.5]
Statistical Analysis 4: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Cytomegalovirus: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 97.1, 95% CI 2-sided [75.5 to 124.8]
Statistical Analysis 5: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Esophageal Candidiasis: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 60.2, 95% CI 2-sided [48.3 to 74.9]
Statistical Analysis 6: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Mycobacterium avium complex: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 98.4, 95% CI 2-sided [70.8 to 136.8]
Statistical Analysis 7: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Cryptococcosis: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 189.5, 95% CI 2-sided [112.3 to 319.5]
Statistical Analysis 8: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Mycobacterium tuberculosis: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 6.2, 95% CI 2-sided [5.2 to 7.4]
Statistical Analysis 9: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Progressive multifocal leukoencephalopathy: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 594.5, 95% CI 2-sided [146.5 to 2411.7]
Statistical Analysis 10: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Lung Candidiasis: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 10.6, 95% CI 2-sided [7.8 to 14.4]
Statistical Analysis 11: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Toxoplasmosis of brain: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 51.5, 95% CI 2-sided [30.3 to 87.5]
Statistical Analysis 12: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Coccidiomycosis: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 6.2, 95% CI 2-sided [3.0 to 12.9]
Statistical Analysis 13: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; Histoplasmosis: Poisson regression models were used to analyze rates of clinical events by HIV and unadjusted incidence rate ratios compared risk in HIV-uninfected persons to HIV-infected persons; Test type: Superiority or Other; p < 0.0001, Poisson Regression; Rate ratio = 13.0, 95% CI 2-sided [7.4 to 23.1]

4. Primary Outcome: Incidence Rate of Liver Failure
Description: Incidence rate of liver failure was calculated as the number of events divided by person-time. Only the first diagnosis of each event per participant was included. Person-time was calculated as the sum of all time contributed by each individual who were KP member from the date of HIV care initiation at that institution or January 1, 1996 for KPNC and January 1, 2000 for KPSC if in care prior to this date. Incidence rate was computed as the number of events per 100,000 person-years.
Time Frame: Up to Week 835
Population: Analysis population included all participants enrolled in the study.
Measure: Number; unit: liver failure per 100,000 person-years
Arm/Group | Cohort 1: HIV Infected | Cohort 2: HIV Uninfected
Number analyzed (Participants) | 24768 | 257600
liver failure per 100,000 person-years | 492 | 105
Statistical Analysis 1: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 4.7, 95% CI 2-sided [4.3 to 5.1]

5. Primary Outcome: Incidence Rate of Liver Related Death
Description: Incidence rate of liver related death was calculated as the number of events divided by person-time. Only the first diagnosis of each event per participant was included. Person-time was calculated as the sum of all time contributed by each individual who were KP member from the date of HIV care initiation at that institution or January 1, 1996 for KPNC and January 1, 2000 for KPSC if in care prior to this date. Incidence rate was computed as the number of events per 100,000 person-years.
Time Frame: Up to Week 835
Population: Analysis population included all participants enrolled in the study.
Measure: Number; unit: death per 100,000 person-years
Arm/Group | Cohort 1: HIV Infected | Cohort 2: HIV Uninfected
Number analyzed (Participants) | 24768 | 257600
death per 100,000 person-years | 202 | 29
Statistical Analysis 1: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 7.0, 95% CI 2-sided [6.0 to 8.2]

6. Primary Outcome: Incidence Rate of Rhabdomyolysis
Description: Incidence rate of Rhabdomyolysis was calculated as the number of events divided by person-time. Only the first diagnosis of each event per participant was included. Person-time was calculated as the sum of all time contributed by each individual who were KP member from the date of HIV care initiation at that institution or January 1, 1996 for KPNC and January 1, 2000 for KPSC if in care prior to this date. Incidence rate was computed as the number of events per 100,000 person-years.
Time Frame: Up to Week 835
Population: Analysis population included all participants enrolled in the study.
Measure: Number; unit: rhabdomyolysis per 100,000 person-years
Arm/Group | Cohort 1: HIV Infected | Cohort 2: HIV Uninfected
Number analyzed (Participants) | 24768 | 257600
rhabdomyolysis per 100,000 person-years | 235 | 28
Statistical Analysis 1: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 8.3, 95% CI 2-sided [7.1 to 9.6]

7. Primary Outcome: Incidence Rate of All-Cause Mortality
Description: Incidence rate of all-cause mortality was calculated as the number of events divided by person-time. Only the first diagnosis of each event per participant was included. Person-time was calculated as the sum of all time contributed by each individual who were KP member from the date of HIV care initiation at that institution or January 1, 1996 for KPNC and January 1, 2000 for KPSC if in care prior to this date. Incidence rate was computed as the number of events per 100,000 person-years.
Time Frame: Up to Week 835
Population: Analysis population included all participants enrolled in the study.
Measure: Number; unit: death per 100,000 person-years
Arm/Group | Cohort 1: HIV Infected | Cohort 2: HIV Uninfected
Number analyzed (Participants) | 24768 | 257600
death per 100,000 person-years | 1827 | 326
Statistical Analysis 1: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 5.6, 95% CI 2-sided [5.3 to 5.9]

8. Primary Outcome: Incidence Rate of Viral Encephalitis
Description: Incidence rate of viral encephalitis (VE) was calculated as the number of events divided by person-time. Only the first diagnosis of each event per participant was included. Person-time was calculated as the sum of all time contributed by each individual who were KP member from the date of HIV care initiation at that institution or January 1, 1996 for KPNC and January 1, 2000 for KPSC if in care prior to this date. Incidence rate was computed as the number of events per 100,000 person-years. The participants with viral encephalitis were followed-up up to 31st December 2009 (730 Weeks).
Time Frame: Up to Week 730
Population: Analysis population included all participants enrolled in the study.
Measure: Number; unit: VE per 100,000 person-years
Arm/Group | Cohort 1: HIV Infected | Cohort 2: HIV Uninfected
Number analyzed (Participants) | 24768 | 257600
VE per 100,000 person-years | 30 | 2
Statistical Analysis 1: Comparison: Cohort 1: HIV Infected vs Cohort 2: HIV Uninfected; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Poisson Regression; Rate ratio = 19.8, 95% CI 2-sided [11.2 to 35.2]

ADVERSE EVENTS:
Description: Due to the retrospective observational nature of study individual adverse events (AEs) were not planned to be collected and reported.
Arm/Group | Cohort 1: HIV Infected | Cohort 2: HIV Uninfected
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Designation of endpoints was based on study team's inputs, as the endpoints were not prioritized in the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.